CLINICAL TRIAL: NCT06850727
Title: A Phase 2a, Two-Part, Open-Label and Randomized Study to Evaluate the Safety and Efficacy of OD-07656 and of Subsequent Vedolizumab Therapy in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: Safety and Efficacy of OD-07656 and of Subsequent Vedolizumab Therapy in Moderately to Severely Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odyssey Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OD-07656-201
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis (UC); UC - Ulcerative Colitis
Keywords: Ulcertative colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- OD-07656 Dosing Regimen 1 (Experimental): Open Label, Oral, twice daily dose
  Interventions: Drug: OD-07656; Drug: Vedolizumab
- OD-07656 Dosing Regimen 2 (Experimental): Randomized, Oral, twice daily dose
  Interventions: Drug: OD-07656; Drug: Vedolizumab
- OD-07656 Dosing Regimen 3 (Experimental): Randomized, Oral, twice daily dose
  Interventions: Drug: OD-07656; Drug: Vedolizumab

INTERVENTIONS:
Drug: OD-07656 — Experimental intervention
Drug: Vedolizumab — Active standard of care comparator

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of OD-07656 in participants with moderately to severely active ulcerative colitis (UC). In addition, the study will evaluate the potential of OD-07656 to enhance the therapeutic benefit of vedolizumab when given after OD-07656.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a confirmed diagnosis of ulcerative colitis (UC)
* Has moderate to severely active UC as defined by the 3-component Modified Mayo clinic score
* Has an inadequate response, loss of response, or intolerance/medical contraindication to at least one of the following therapies: oral aminosalicylates, corticosteroids, immunosuppressants, anti-tumor necrosis factor biologic, anti-interleukin 12/23 biologic, Janus kinase inhibitors, or sphingosine-1-phosphate (S1P) modulators

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has diagnosis of Crohn's disease or indeterminate colitis
* Has had extensive colonic resection
* Has colostomy or ileostomy
* Has uncontrolled primary sclerosing cholangitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in 3-component modified Mayo Clinic Score (MMCS) from baseline to after treatment with OD-07656 | Baseline and 12 weeks
  The 3-component MMCS ranges from 0 to 9 and is composed of endoscopic assessment, rectal bleeding and stool frequency subscores with each of the components ranging from 0 to 3, with higher scores indicating more severe disease.
Incidence of treatment-emergent adverse events (TEAEs) and treatment discontinuations due to TEAEs with OD-07656 treatment | Up to 12 weeks

SECONDARY OUTCOMES:
Proportion of participants who achieve clinical remission | Baseline and 12 weeks
  Clinical remission is based on the MMCS and is defined as endoscopic subscore of 0 or 1, rectal bleeding subscore of 0 and stool frequency subscore of 0 or 1 and not greater than baseline.
Proportion of participants who achieve clinical remission with vedolizumab treatment, following OD-07656 treatment | Baseline and 50 weeks
  Clinical remission is based on the MMCS and is defined as endoscopic subscore of 0 or 1, rectal bleeding subscore of 0 and stool frequency scubscore of 0 or 1 and not greater than baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Odyssey Therapeutics
Locations (32):
- Australia (6):
  - Sunshine Coast University, Birtinya
  - Eastern Health, Box Hill
  - Coastal Digestive Health, Maroochydore
  - Alfred Health, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Royal Melbourne Hospital, Parkville
- Medical University of Graz, Graz, Austria
- Canada (2):
  - CHUM, Montreal
  - Montreal General Hospital/McGill University, Montreal
- CHUM - Pavillon R, Polička, Czechia
- Jordan (3):
  - Jordan University Hospital, Amman
  - The Specialty Hospital (TSH) / Advanced Clinical Center, Amman
  - Irbid Specialty Hospital, Irbid
- The Hospital of Lithuanian University of Health Sciences, Kaunas, Lithuania
- IMSP Spitalul Clinic Republican Timofei Moneaga, Chisinau, Moldova
- New Zealand (5):
  - PCRN Auckland, Auckland
  - PCRN Christchurch, Christchurch
  - PCRN Waikato, Hamilton
  - PCRN Tasman, Nelson
  - PCRN Wellington, Upper Hutt
- Poland (8):
  - Centrum Medyczne, Bydgoszcz
  - Centrum Medyczne LukaMed, Chojnice
  - Vita Longa Sp. z.o.o., Katowice
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia Sp. z.o.o, Sopot
  - Nowe zdrowie-CK, Kiełtucki, Staszów
  - Medical Network Company, Warsaw
  - Penta Hospitals Przychodnie, Wroclaw
- Ukraine (4):
  - Regional Clinical Hospital, Ivano-Frankivsk
  - Medical centre of ARENSIA Exploratory Medicine LCC, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv
  - Lviv Regional Clinical Hospital, Lviv

IPD SHARING:
Plan to Share IPD: Undecided